CLINICAL TRIAL: NCT05720273
Title: The Effect of Neutrophil Gelatinase-associated Lipocalin Derived From Osteoblasts and Vascular Smooth Muscle Cells on Vascular Calcification in Chronic Kidney Desease and the Intervention of Paliscalcitol - Clinical Research Section
Brief Title: Neutrophil Gelatinase-associated Lipocalin VS Vascular Calcification in Maintenance Hemodialysis Patients
Acronym: NGAL
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Xiaoyan Jia (Other)
Responsible Party: Sponsor-Investigator, Xiaoyan Jia, Clinical Professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: YXLL-KY-2022(066)
Record Dates: First submitted 2022-11-10; First posted 2023-02-09 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Chronic Kidney Disease-Mineral and Bone Disorder
Keywords: Chronic Kidney Disease-Mineral and Bone Disorder; Calcitriol Receptor; Lipocalin-2; Vascular Calcification
MeSH Terms: conditions — Chronic Kidney Disease-Mineral and Bone Disorder; Vascular Calcification | interventions — Calcitriol

STUDY DESIGN:
Intervention Model Description: Maintenance hemodialysis patients with secondary hyperparathyroidism
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Palicalcitol (Experimental): Maintenance hemodialysis patients with secondary hyperparathyroidism (SHPT) treat with palicalcitol
  Interventions: Drug: palicalcitol

INTERVENTIONS:
Drug: palicalcitol — This study does not interfere with the clinical medication of the researchers, and the usage and dosage of the drugs will be recorded according to the actual use. The recommended starting dose of palicalcitol may be based on body weight, baseline iPTH, or combined with prior medication. Dose adjustment should be determined according to pre-dialysis iPTH, Ca and P. iPTH levels should be maintained at 150-300pg/ml, while Ca and P levels should be closely monitored. If hypercalcemia occurs, the dose should be reduced or medication should be discontinued until these parameters return to normal; Subsequently, the dose of palicalcitol should be restarted at a lower dose. If PTH levels decrease as a result of treatment, the dose of medication may need to be reduced accordingly. The dose adjustment interval is 2-4 weeks, and the dose can be adjusted immediately for safety reasons.
  Other Names: Calcitriol; Calcimimetics

SUMMARY:
The goal of this observational study or clinical trial is to learn about the effect of neutrophil gelatinase-associated lipocalin (NGAL) on vascular calcification in maintenance hemodialysis patients with secondary hyperparathyroidism (SHPT). The main question it aims to answer is: the predictive effects of blood NGAL level on the efficacy of palicalcitol in the treatment of SHPT and the adverse reactions of vascular calcification progression. Participants will be treated with palicalcitol, followed up and undergo routine series of Chronic Kidney Disease-Mineral and Bone Disorder associated tests before and after treatment.

DETAILED DESCRIPTION:
1. Sample size calculation: Because there was no previous study on the change of blood NGAL level in MHD patients with palicalcitol; refer to the NGAL changes before and after parathyroidectomy :N=12 NGAL715.84(578.73, 988.14)ng/mL before and 688.42(660.00, 760.26)ng/mL 4-7 days after surgery (p=0.071, paired T-test). According to the 20% loss rate; The sample size is finally determined to be 80 cases.
2. Patients: maintenance hemodialysis patients with secondary hyperparathyroidism (SHPT).
3. Palicalcitol injection
4. Follow-up The patients are followed up for 1 year.
5. Statistical methods All statistical tests are conducted by two-sided test, and the first type of error is 0.05 (α value) to determine the statistical significance of the difference. Quantitative data includ efficacy, laboratory test indicators, such as the number of cases, mean, median, standard deviation and range description. Qualitative data includ comorbidities, described in terms of frequency, composition or percentage. Statistical test: The parameter test method is preferred. If the data distribution differs greatly from the requirements of testing the hypothesis, the non-parameter test method will be used. Patients will be divided into two groups according to circulating NGAL levels before treatment; the clinical characteristics, changes of NGAL level, the efficacy of palicalcitol (changes of iPTH) and the main adverse reactions (increased blood calcium and phosphorus, progress of vascular calcification) are compared between two groups. T test or rank sum test are used for difference test. The correlation between blood NGAL level, VC score and CKD-MBD assay indexes is analyzed by pair-wise correlation and logistic multivariate regression.

ELIGIBILITY:
Inclusion criteria:

* Chronic kidney disease (CKD) maintenance hemodialysis patients with secondary hyperparathyroidism (SHPT), iPTH>300pg/ml
* Age 18-65 years old
* Haven't used anti-PTH agents within 3 months
* Signed informed consent

Exclusion criteria:

* Allergic to vitamin D or similar drugs
* Vitamin D poisoning
* Expected survival is less than one year
* Acute inflammations, active liver disease, tumor, hospitalization within 3 months
* Fractures, major trauma or operations within 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline plasma NGAL levels at 12months | 12months
  Elisa

SECONDARY OUTCOMES:
Change from baseline vascular calcification at 12months | 12months
  Coronary calcification scores (CACS) from serial computed tomographic images with the Agatston method is used to evaluate cardio-vascular calcification, 1 point=130~199HU；2 points=200~299HU；3 points =300~399HU；4 points≥400HU. Abdominal aortic calcification score (AACS) is measured by Kauppila method from lateral dual-energy X-ray absorptiometry spine, 0-3 points. Anterior chest radiographs is used to perform simple calcification scores for aortic arch knob, 0-100%. Higher scores mean a worse outcome.

OTHER OUTCOMES:
Change from baseline Chronic Kidney Disease-Mineral and Bone Disorder associated laboratory tests at 12months | 12months
  Serum calcium and phosphorus are analyzed by Beckman automatic biochemical analyzer in our laboratory center. Blood iPTH measured by ELISA.
Change from baseline bone density tests at 12months | 12months
  Quantitative computed tomography (QCT) measurements are performed at the lumbar spine (mean of L 1 and L 2 entire vertebral bodies, excluding posterior processes) and hip.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-04-10): https://cdn.clinicaltrials.gov/large-docs/73/NCT05720273/ICF_000.pdf